CLINICAL TRIAL: NCT03037684
Title: Selective Activation of Unmyelinated Skin Nerve Fibres Using Slow Depolarising Transcutaneous Electrical Stimulation in Patients With Neuropathic Pain or Chronic Postoperative Pain
Brief Title: Depolarising Electrical Skin Stimulation in Neuropathic and Postoperative Pain
Status: Recruiting | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2016-15
Record Dates: First submitted 2017-01-16; First posted 2017-01-31 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Neuropathy;Peripheral
Keywords: neuropathic pain; chronic postoperative pain
MeSH Terms: conditions — Neuritis; Neuralgia; Pain, Postoperative | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic pain: individuals suffering from chronic pain
  Interventions: Diagnostic Test: neurophysiology
- neuropathic pain: individuals suffering from neuropathic pain
  Interventions: Diagnostic Test: neurophysiology

INTERVENTIONS:
Diagnostic Test: neurophysiology — electrophysiologic measurements of peripheral nerves

SUMMARY:
The aim of the study is to evaluate voltage gated sodium channel (NaV1.7) dependent pain phenomena in neuropathic pain and chronic postoperative pain.

DETAILED DESCRIPTION:
Sinus-like electrical stimulation may depolarize unmyelinated skin nociceptors involving NaV1.7 channels. In this case electrical stimulation may provoke pain already with very low currency intensity which normally not provoke pain in healthy subjects. This may be predictive for pain relief due to the sodium channel blocker lidocaine 5% patch.

The study will characterize pain states in peripheral neuropathic pain as well as within the painful scar in chronic postoperative pain with regard to the involvement of NaV1.7 channels.

In addition, the pain site in chronic postoperative pain (scar) will be characterized by laser-evoked potentials (LEP) and quantitative sensory testing (QST).

Pain related questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Group (1) patients with neuropathic pain
* Group (2) patients with chronic postoperative pain

Exclusion Criteria (both Groups):

* severe psychiatric disorder requiring hospitalisation in the past
* any neurological disease other than the pain diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with neuropathic pain or with chronic postoperative pain
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | at baseline and during electric nerve stimulation
  numeric rating scale (NRS), rating from 0-10, 0=no pain, 10=maximum pain imaginable

SECONDARY OUTCOMES:
heat pain threshold | baseline
  Ramped stimuli (+1 degree Celsius / sec) that are terminated when the subject presses a button.
cold pain threshold | baseline
  Ramped stimuli (-1 degree Celsius / sec) that are terminated when the subject presses a button.
mechanical detection threshold | baseline
  Fine plastic hairs with different bending forces are applied to the skin to determine the mechanical detection threshold.
mechanical pain threshold | baseline
  Differently weighted pinprick stimuli are applied at a rate of 2sec on and 2sec off in an ascending order until the first percept of sharpness is reached.
mechanical pain sensitivity | baseline
  Differently weighted pinprick stimuli are applied to obtain a stimulus- response function for pinprick-evoked pain. Subjects were asked to give a pain rating for each stimulus (rating from 0-10, 0=no pain, 10=maximum pain)
dynamic mechanical allodynia | baseline
  Different stimuli, tactile and pinprick are applied with the subject giving numerical pain ratings for each stimulus (rating from 0-10, 0=no pain, maximum pain).
vibration detection threshold | baseline
  Tuning fork is placed over a bony prominence until the subject cannot not feel vibration any more.
pressure pain threshold | baseline
  A pressure gauge that exerts forces of ascending stimulus intensities is applied as a slowly increasing ramp over a muscle.
LEP latency | baseline
  latency of N2 and P2 components of laser evoked potential signal curve
LEP amplitude | baseline
  amplitude of laser evoked potential signal curve
stadium of pain chronification | baseline
  assessment of the stadium of pain chronification (stadium 1-3) using standardized questionnaire
pain severity | baseline
  assessment of pain severity (grade 1-4) using the Chronic Pain Grading Questionnaire
physical health status | baseline
  assessing the physical health status using the Short Form-12 questionnaire
mental health status | baseline
  assessing the mental health status using the Short Form-12 questionnaire
anxiety | baseline
  assessing anxiety using the Hospital Anxiety and Depression Scale questionnaire
depression | baseline
  assessing Depression using the Hospital Anxiety and Depression Scale questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Pain Medicine, Nottwil, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110